CLINICAL TRIAL: NCT04163744
Title: Effectiveness and Safety of Induction of Labour Using a Double Balloon Catheter (INDOBA)
Acronym: INDOBA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-CRB-2019-70
Record Dates: First submitted 2019-11-12; First posted 2019-11-15 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Induction of Labour
Keywords: Induction of labour; Double balloon catheter; Vaginal delivery rate; Mechanical method; in-patient; out-patient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Double balloon catheter — Induction of labour with double balloon catheter

SUMMARY:
The goal of induction of labor is to achieve vaginal delivery by stimulating uterine contractions before the spontaneous onset of labor. Generally, induction of labor has merit as a therapeutic option when the benefits of expeditious delivery outweigh the risks of continuing the pregnancy.

The first part of this process is called cervical ripening. The goal is to facilitate the process of cervical softening, thinning, and dilating with resultant reduction in the rate of failed induction and induction to delivery time. Cervical remodeling is a critical component of normal parturition.

Effective methods for cervical ripening include the use of mechanical and pharmacological methods.

There are many induction methods: pharmacological and mechanical.

Nowadays, induction of labour is one of the most frequent obstetric interventions, performed in 25% of pregnancies. Generally, better maternal and neonatal outcomes are achieved if the risks of continuing pregnancy outweigh the benefits.

Cervical ripening is the first part of the induction process, which consists in relaxing and softening the uterine cervix prior to the onset of uterine dynamics.

For this purpose, there are available pharmacological (mainly prostaglandin) and mechanical methods (including the balloon probes: Foley catheter or double cervical balloon). Despite being equally effective in vaginal delivery and caesarean section rate, there has been registered an increased risk of uterine hyperdynamic with the use of prostaglandin in contrast to the use of balloon probes, which may lead to an increased risk of fetal distress.

Concerning balloon probes, various published studies conclude that it is an effective and safe cervical ripening method, without increasing the risk of maternal infection (chorioamnionitis / endometritis) or neonatal infection.

The use of balloon probes could be established as first-choice method of induction of labour, reducing the risk of uterine hyperdynamic and the likelihood of intrauterine fetal distress derived from the use of prostaglandin.

The balloon probe safety makes it an ideal method for performing cervical ripening at home (out-patient) in low-risk pregnancies, increasing the satisfaction of women who desire it and reducing the economic cost for the hospital.

The purpose of this study is to assess the effectiveness and safety of double balloon catheter (CRB-Cook®) in induction of labour.

The main objective is to provide evidence that there are no differences in caesarean section rate between induction of labour performed with Cook double balloon catheter in out-patient and in-patient compared with a cohort of induction of labour with pharmacological methods (dinoprostone and misoprostol).

Two clinical studies will be carried out for this purpose:

1. Prospective cohort observational study
2. Historical case-control study

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* Age: ≧ 18 years
* Ability to read and understand informed consent
* Unique or multiple pregnancies (monochorionic or dichorionic twins)
* ≧37 weeks of pregnancy
* Unfavourable cervix (Bishop test: < 7)

Exclusion Criteria:

* >2 foetus pregnancies
* < 37 or ≧42 weeks of pregnancy
* Prelabour rupture of membranes
* Vaginal delivery contraindication

  * Placenta previa (occlusive and not occlusive)
  * Vasa previa
  * Transverse or oblique lie
  * Umbilical cord procubitus or prolapse
  * Corporal uterine surgery with entrance into the uterine cavity
  * Antecedent of ≧ 2 caesarean section
  * Antecedent of inverted T caesarean section
  * Antecedent of uterine rupture
  * Active genital herpes infection
  * Cervical carcinoma
  * Severe maternal pathology
* Breech lie
* ≥ 7 Bishop score
* Non-reassuring fetal cardiotocographic registration
* Indication of immediate delivery
* Stillbirth of malformed foetus

Also, patients to be included in the out-patient group should comply with the following criteria:

Inclusion criteria:

* Low-risk pregnancies
* ≤ 2 previous deliveries
* Patient acceptation and good comprehension of the instructions
* Maximum 30 minutes of distance to the hospital.
* Possibility of telephone communication at any moment
* To be accompanied by someone during the entire process at home

Exclusion criteria:

- Positive screening for vaginal / rectum group B streptococcal infection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-10-10 (Actual); Primary Completion 2020-11-01 (Estimated); Study Completion 2021-02-02 (Estimated)

PRIMARY OUTCOMES:
Effectiveness Vaginal delivery / caesarean section rate | 12 months
  Measure vaginal delivery and caesarean rate of induction of labour with double balloon catheter

SECONDARY OUTCOMES:
Safety of patient and foetus | 12 months
  Measured through complications and adverse effects registered during induction of labour
Patients satisfaction | 12 months
  Measured as global satisfaction with the use of double balloon catheter as induction of labour method with an analog visual scale from 0 to 10

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Llurba, MD, PhD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

REFERENCES:
- [Result] WHO recommendations: Induction of labour at or beyond term. Geneva: World Health Organization; 2018. Available from http://www.ncbi.nlm.nih.gov/books/NBK535795/ PMID 30629393
- [Result] Chen W, Xue J, Peprah MK, Wen SW, Walker M, Gao Y, Tang Y. A systematic review and network meta-analysis comparing the use of Foley catheters, misoprostol, and dinoprostone for cervical ripening in the induction of labour. BJOG. 2016 Feb;123(3):346-54. doi: 10.1111/1471-0528.13456. Epub 2015 Nov 5. PMID 26538408
- [Result] Ten Eikelder ML, Mast K, van der Velden A, Bloemenkamp KW, Mol BW. Induction of Labor Using a Foley Catheter or Misoprostol: A Systematic Review and Meta-analysis. Obstet Gynecol Surv. 2016 Oct;71(10):620-630. doi: 10.1097/OGX.0000000000000361. PMID 27770132
- [Result] Diederen M, Gommers J, Wilkinson C, Turnbull D, Mol B. Safety of the balloon catheter for cervical ripening in outpatient care: complications during the period from insertion to expulsion of a balloon catheter in the process of labour induction: a systematic review. BJOG. 2018 Aug;125(9):1086-1095. doi: 10.1111/1471-0528.15047. Epub 2018 Jan 10. PMID 29211328
- [Result] Vaknin Z, Kurzweil Y, Sherman D. Foley catheter balloon vs locally applied prostaglandins for cervical ripening and labor induction: a systematic review and metaanalysis. Am J Obstet Gynecol. 2010 Nov;203(5):418-29. doi: 10.1016/j.ajog.2010.04.038. PMID 20605133
- [Result] McMaster K, Sanchez-Ramos L, Kaunitz AM. Evaluation of a Transcervical Foley Catheter as a Source of Infection: A Systematic Review and Meta-analysis. Obstet Gynecol. 2015 Sep;126(3):539-551. doi: 10.1097/AOG.0000000000001002. PMID 26244535
- See also: Related Info — http://www.nice.org.uk/guidance/ipg528/resources/insertion-of-a-double-balloon-catheter-for-induction-of-labour-in-pregnant-women-without-previous-caesarean-section-pdf-1899871812579013